CLINICAL TRIAL: NCT01872884
Title: Sedation Versus General Anesthesia for Endovascular Therapy in Acute Stroke - Impact on Neurological Outcome
Acronym: ANSTROKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Alexandros Rentzos, MD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ANSTROKE; ALFGBG-75870 (Other Grant/Funding Number: Swedish State Support for Clinical Research (ALFGBG-75870))
Record Dates: First submitted 2013-06-04; First posted 2013-06-07 (Estimated); Last update posted 2017-10-11 (Actual); Status verified 2017-10

CONDITIONS: Ischemic Stroke
Keywords: Stroke; Ischemic stroke; Acute stroke; Embolectomy; Endovascular therapy; Intra-arterial therapy; Sedation; Anesthesia
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Intubation, Intratracheal; Remifentanil; Conscious Sedation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- General anaesthesia (Experimental): General anaesthesia with mechanical ventilation. Sevorane Remifentanil. Bloodpressure control, systolic pressure 140-180 mmHg.
  Interventions: Drug: Sevorane Remifentanil
- Sedation (Placebo Comparator): Sedation with spontaneous breathing. Remifentanil. Bloodpressure control, systolic pressure 140-180 mmHg
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Sevorane Remifentanil — Sevorane Remifentanil
  Other Names: tracheal intubation
  Arms: General anaesthesia
Drug: Remifentanil — Remifentanil
  Other Names: Conscious sedation
  Arms: Sedation

SUMMARY:
The purpose of this study is to evaluate whether general anesthesia or sedation technique is preferable during embolectomy for stroke, measured in terms of three months neurological impairment. In addition we study if there is any difference between the methods regarding complication frequency.

DETAILED DESCRIPTION:
Stroke is a common cause of neurological disability. Early diagnosis of ischemic stroke now enables treatment with thrombolysis and / or endovascular therapy (embolectomy). In order to implement this procedure, the duration of which varies from 2-6 hours, the patient has to remain immobilized. Two techniques are currently used routinely to achieve this.

One technique is general anaesthesia, that will ensure that the patient is completely immobile throughout the procedure, which is an advantage from a neuroimaging perspective. A disadvantage is that preparation for, and the induction of anesthesia prolongs the time to embolectomy. Another disadvantage may be that the patient´s blood pressure drops during anesthesia, which could impair the brain blood supply and subsequently neurological outcome. The ability to evaluate the patient's neurological symptoms also disappears.

The second technique consists of sedation during surgery. The advantages of this technique are that the time to the beginning of embolectomy is getting shorter and the blood pressure becomes more stable. One drawback is that it cannot guarantee that the patient remains immobile throughout the procedure, which increases the risk of motion artifacts and may lead to the duration of embolectomy becomes prolonged. There is also a risk of hypoventilation and the patient aspirates during surgery.

Retrospective studies suggest that patients receiving general anesthesia have worse neurologic outcome three months after stroke. This could be explained by more or less pronounced anesthesia-induced episodes of hypotension, compared with lightly sedated patients with more stable blood pressure. In these retrospective analyzes, however, the patients who received general anesthesia were, neurologically speaking, more ill than patients who only received sedation. This may probably, at least in part, explain why anesthetized patients have a worse neurologic outcome. In these retrospective studies, many centers were involved, with various endovascular and anesthesia procedures.

ELIGIBILITY:
Inclusion Criteria:Patients with acute stroke considered for thrombectomy and meeting the following inclusion criteria included:

1. the patient is ≥ 18 years
2. the patient has a CT angio verified embolization * and / or a NIHSS scores ** ≥ 10 (R) or 14 (L) depending on the side engagement
3. embolectomy (= groin puncture) started <8 hours after symptom onset

   * Embolus in one of the following arteries: internal carotid artery, anterior cerebral (A1 segment), cerebri media (M1 segment) and proximal cerebri media branches (M2 segment).

     * NIHSS (National Institutes of Health Stroke Scale). Patients with embolus in left hemisphere circulation require ≥ 14 points, while patients with embolus in the right hemisphere circulation require ≥ 10 points. This is because occlusion on the right side does not usually cause aphasia, a symptom that usually leads to higher total score of NIHSS.

Exclusion Criteria:

1. the patient must receive general anesthesia, for medical reasons, according to the responsible anesthesiologist
2. the patient cannot receive general anesthesia, for medical reasons, according to the responsible anesthesiologist
3. the patient has an embolization of posterior brain vessels
4. CT-confirmed intracerebral hemorrhage
5. spontaneous recanalization or spontaneous neurological improvement
6. any other reason that does not allow embolectomy (co-morbidities)
7. premorbid MRS ≥ 4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2013-11-14 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Neurological outcome in the two different arms | 90 days
  Neurological outcome is measured as modified Rankin Scale (mRS), 90d post stroke.

SECONDARY OUTCOMES:
NIHSS(National Institutes of Health Stroke Scale) | Day 3,7,90
  Change in NIHSS score on day 3, day 7 and 3 months compared to admission to hospital
The degree of recanalization and reperfusion | 1 day (After completed embolectomy)
  Measures as modified TICI(Thrombolysis In Cerebral Infarction)score
Periprocedural complications | Perioperatively
Infarction magnitude | Day 1 to Day 90
  CT (computer tomography scan) Day 1 incl CTperfusion MR (magnetic resonance imaging) on day 3 (2-4) and 3 months Brain damage markers (GFAP, Tau, S-100B) before, 2, 24, 48, 72 hours and 3 months after the procedure.
Quantitative EEG changes | Day 1,2,90
  Quantitative EEG (electro encephalography) days 1, 2, and three months after onset
Time consumption | Periprocedural
  Time consumed from: stroke onset to CT angiography, CT angiography to start of anesthesia / sedation, stroke onset to start of embolectomy and duration of embolectomy.
Hospital length of stay | Approximately 7-14 days
  Hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Alexandros Rentzos, MD, Principal Investigator — Diagnostic and interventional Neuroradiology, Radiology department, Sahlgrenska Academy, University of Gothenburg; Pia Löwhagen Henden, MD, Principal Investigator — Anesthesiology, Sahlgrenska Academy, University of Gothenburg; Sven-Erik Ricksten, MD PhD Prof, Study Director — Sahlgrenska Academy, University of Gothenburg
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jumaa MA, Zhang F, Ruiz-Ares G, Gelzinis T, Malik AM, Aleu A, Oakley JI, Jankowitz B, Lin R, Reddy V, Zaidi SF, Hammer MD, Wechsler LR, Horowitz M, Jovin TG. Comparison of safety and clinical and radiographic outcomes in endovascular acute stroke therapy for proximal middle cerebral artery occlusion with intubation and general anesthesia versus the nonintubated state. Stroke. 2010 Jun;41(6):1180-4. doi: 10.1161/STROKEAHA.109.574194. Epub 2010 Apr 29. PMID 20431082
- [Background] Nichols C, Carrozzella J, Yeatts S, Tomsick T, Broderick J, Khatri P. Is periprocedural sedation during acute stroke therapy associated with poorer functional outcomes? J Neurointerv Surg. 2010 Mar;2(1):67-70. doi: 10.1136/jnis.2009.001768. Epub 2009 Dec 17. PMID 20431708
- [Background] Abou-Chebl A, Lin R, Hussain MS, Jovin TG, Levy EI, Liebeskind DS, Yoo AJ, Hsu DP, Rymer MM, Tayal AH, Zaidat OO, Natarajan SK, Nogueira RG, Nanda A, Tian M, Hao Q, Kalia JS, Nguyen TN, Chen M, Gupta R. Conscious sedation versus general anesthesia during endovascular therapy for acute anterior circulation stroke: preliminary results from a retrospective, multicenter study. Stroke. 2010 Jun;41(6):1175-9. doi: 10.1161/STROKEAHA.109.574129. Epub 2010 Apr 15. PMID 20395617
- [Background] Davis MJ, Menon BK, Baghirzada LB, Campos-Herrera CR, Goyal M, Hill MD, Archer DP; Calgary Stroke Program. Anesthetic management and outcome in patients during endovascular therapy for acute stroke. Anesthesiology. 2012 Feb;116(2):396-405. doi: 10.1097/ALN.0b013e318242a5d2. PMID 22222475
- [Derived] Tosello R, Riera R, Tosello G, Clezar CN, Amorim JE, Vasconcelos V, Joao BB, Flumignan RL. Type of anaesthesia for acute ischaemic stroke endovascular treatment. Cochrane Database Syst Rev. 2022 Jul 20;7(7):CD013690. doi: 10.1002/14651858.CD013690.pub2. PMID 35857365
- [Derived] Lowhagen Henden P, Rentzos A, Karlsson JE, Rosengren L, Leiram B, Sundeman H, Dunker D, Schnabel K, Wikholm G, Hellstrom M, Ricksten SE. General Anesthesia Versus Conscious Sedation for Endovascular Treatment of Acute Ischemic Stroke: The AnStroke Trial (Anesthesia During Stroke). Stroke. 2017 Jun;48(6):1601-1607. doi: 10.1161/STROKEAHA.117.016554. PMID 28522637